CLINICAL TRIAL: NCT05034666
Title: Endotracheal Tube Cuff Inflation Pressure Varieties and Response to Education Among Anesthetists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: ETT cuff pressure
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Endotracheal Tube

STUDY DESIGN:
Intervention Model Description: anaesthetists of anaesthesia department on Suez canal university
Who Masked: Participant
Masking Description: the participants are not informed about the visit, and the investigator is measuring the ETT cuff pressure in the absence of the participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before education (Active Comparator): Before alarming the participant anaesthetists about the pressure values of their practice in inflating the ETT cuff.
  This is before applying the intervention which is informing and educating the participant anaesthetists about the proper ETT cuff pressure.
  Interventions: Behavioral: Before the education program
- After education (Active Comparator): After alarming the participant anaesthetists about the pressure values of their practice in inflating the ETT cuff.
  This is after applying the intervention which is informing and educating the participant anaesthetists about the proper ETT cuff pressure.
  Interventions: Behavioral: After the education program

INTERVENTIONS:
Behavioral: Before the education program — Before applying the education program of the endotracheal cuff pressure inflation to the participating anaesthetists.
  Arms: Before education
Behavioral: After the education program — After applying the education program of the endotracheal cuff pressure inflation to the participating anaesthetists.
  Arms: After education

SUMMARY:
Cuff pressure is essential in endotracheal tube management. Guidelines recommend a cuff pressure of 20 to 30 cm H2O. One study, for instance, found that cuff pressure exceeded 40 cm H2O in 40-to-90% of tested patients.

This study will investigate the endotracheal ETT cuff inflation pressure applied by the participating anaesthetists, and their response after being informed about the pressure the participants will apply.

DETAILED DESCRIPTION:
Although the increasing uses of different supraglottic devices as an alternative, the traditional endotracheal intubation is still considered the commonly used method for managing the airway of a generally anaesthetized patient. After passing the endotracheal tube through the larynx, the anaesthetist inflates the cuff or asks the anaesthesia technician to inflate it. How much air is injected into the cuff is not a major concern for almost all anaesthetists and they usually depend on palpating the external cuff tense to judge is it too much, accurate or not enough? Cuff pressure is essential in endotracheal tube management. Guidelines recommend a cuff pressure of 20 to 30 cm H2O. Inflation of the cuff of pressure more than 30 cm H2O can damage the tracheal mucosa by compromising capillary perfusion. When pressures are greater than 50 cm H2O, total obstruction of tracheal blood flow occurs. For long times, without any evidence-based data, it has been believed that well-trained anaesthetists are capable of determining proper ETT cuff pressures. It is presumed that anaesthetists can detect appropriate inflation pressure and overinflated ETT cuff by palpating the ETT pilot balloon. Adequacy of cuff inflation is conventionally determined by palpation of the external balloon. Previous studies suggest that this approach is unreliable. One study, for instance, found that cuff pressure exceeded 40 cm H2O in 40-to-90% of tested patients. However, increased awareness of over-inflation risks may have improved recent clinical practice.

The aim of the work: This study will investigate the endotracheal cuff inflation pressure applied by the participating anaesthetists, and their response after being informed about the pressure the participants will apply. Material and Methods: Type of the study: Prospective controlled single-blind study. Settings: After obtaining approval by the Ethics Committee of the Suez Canal University Hospital, and written informed consent with an explanation regarding the purpose, effects, technique, and complications, all anaesthetists, working currently in the facility, are included.

ELIGIBILITY:
Inclusion Criteria:

* anaesthetists
* works at Suez canal university hospital
* resident, registrar, or senior registrar

Exclusion Criteria:

* refusal to participate
* who will not complete the 2 rounds 3 readings each

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
accuracy in inflating the cuff of the endotracheal tubes | immediately after fixation of the endotracheal tube during general anaethesia
  assessment of the Anesthetists' accuracy in inflating the cuff of the endotracheal tubes used to maintain the airway of generally anaesthetized patients the change following feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided